CLINICAL TRIAL: NCT01063673
Title: The Relation Between Running Patterns and Overuse Injuries in Runners
Status: Completed | Type: Observational
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Collaborators: University of Aarhus (Other); Bispebjerg Hospital (Other); Foot and Ankle Research Northern Denmark (Unknown)
Responsible Party: Sponsor
Other Study IDs: M-20110114
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Overuse Injuries
Keywords: Running, overuse injury, limits humans
MeSH Terms: conditions — Cumulative Trauma Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Active runners: Observational follow-up study on 39 runners

SUMMARY:
Running patterns are thought to have a major influence on the development of Running Related Injuries (RRI), however to studies have documented such relationship. Thus, the aim of the study is to investigate the association between running patterns and overuse injuries in runners.

DETAILED DESCRIPTION:
Running patterns are thought to have a major influence on the development of Running Related Injuries (RRI).

Worldwide, running is a sport practiced by many individuals to improve cardio-respiratory function, health and well-being. Although running positively contributes to health, there is also a risk of running related injuries (RRI). At best, the consequence of RRI´s is a periodic absence from physical activity, with the athlete returning to sport within weeks. In the worst case, the injury is a chronic painful condition, causing a sedentary lifestyle without physical activity. This is undesirable since physical inactivity increases the risk of lifestyle diseases and death.

In Denmark it is estimated that 4.500 deaths each year can be attributed directly to inactivity. Furthermore, inactivity leads to reduced quality of life compared to active persons. To avoid people getting a sedentary lifestyle prevention of RRI are necessary.

To define a prevention strategy, one must have knowledge about risk factors and causation. Many risk factors have been proposed. Among these, running patterns and foot type are thought to play a major role in the development of RRI. However, very few firm conclusions can be made based on the existing literature, often because of methodical problems. Consequently, it is suggested to design large scale prospective studies controlling for multiple variables. Furthermore, studies should differentiate between novice, elite and extreme runners. Thus, the study design in this project will take these suggestions into account.

The aim of the study is to investigate the association between running patterns and overuse injuries in runners.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 65 years old
* has a GPS-watch that can measure training data (Garmin Forerunner 205,305 or 405)
* has registered their training (if they have run) for a period of at least three months before the inclusion in the trial
* has an e-mail address

Exclusion Criteria:

* does not wish to keep a training diary
* has not registered training data in the follow-up period
* has had an injury in the leg within the last three months before baseline
* active with another tough sports, cf. American College of Sports Medicine
* psychic condition that does not allow participation
* cannot read or understand Danish

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Beginners: n = 1000. By means of the Danish Personal Register adult citizens (age 18-65 years) from Aarhus Municipality are identified, contacted by phone, and invited to participate in the study. A question on running experience in the past is used to assess the novelty to running. 500 beginners with previous running experience and 500 beginners without previous running experience (former runners) will be included in the study. It is estimated that 11000 persons have to be contracted to include 1000 individuals. Healthy persons who have not sustained an injury in the lower extremity in the last 3 months before inclusion and who have not been running for the last 12 months, are eligible for the study. Participants are excluded if there are absolute contraindications for vigorous physical activities according to the ACSM, or in case of unwillingness to keep a training log / wear a heart rate belt during training.
Sampling Method: Non-Probability Sample
Enrollment: 940 (Actual)
Dates: Start 2010-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Injury defined as any musculoskeletal complaint of the lower extremity or back causing a restriction of running for at least 1 week. | a two-week period before the injury arises

CONTACTS AND LOCATIONS:
Overall Officials: Sten Rasmussen, M.D., DrMSc, Principal Investigator — Orthopaedic Division, North Denmark Region, Aalborg Hospital - Aarhus University Hospital, Denmark
Locations (2):
- Denmark (2):
  - Northern Orthopaedic Division, Aalborg University Hospital, Aalborg, Northern Jutland
  - VIA UC, Holstebro